CLINICAL TRIAL: NCT05191745
Title: Long-acting Parasternal Blocks for Analgesia After Cardiac Surgery: A Randomized, Controlled, Double-Blinded Clinical Trial
Brief Title: Long-acting Parasternal Blocks for Analgesia After Cardiac Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Matthew Cameron, Assistant Professor, Jewish General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2022-3125
Record Dates: First submitted 2021-12-03; First posted 2022-01-13 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Coronary Artery Bypass Graft Surgery
Keywords: Cardiac surgery; Pain
MeSH Terms: conditions — Pain | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Patients will receive bilateral parasternal blocks at the end of cardiac surgery.
  Interventions: Drug: Parasternal blocks
- Control group (Placebo Comparator): Patients will receive all standard care as per the hospital protocols.
  Interventions: Drug: Standard of care

INTERVENTIONS:
Drug: Parasternal blocks — Parasternal block with Bupivacaine 0.25% + Epinephrine 1:200,000 x 60cc + Dexamethasone 5mg and Dexmedetomidine 50mcg
  Other Names: pecto-intercostal fascial blocks
  Arms: Intervention group
Drug: Standard of care — All standard management of postoperative pain, as per local protocols
  Arms: Control group

SUMMARY:
This is a randomized, double-blind, controlled clinical trial is to evaluate the duration of efficacy of parasternal blocks with the use of local anesthetic adjuncts for analgesia after coronary artery bypass grafting surgery.

DETAILED DESCRIPTION:
This study will randomize patients to either standard pain control protocols or parasternal blocks after coronary artery bypass grafting-only surgery. This study will specifically examine the effectiveness and duration of analgesia of parasternal blocks with local anesthetic adjuncts, Dexamethasone 10mg and Dexmedetomidine 50mcg, added to the local anesthetic mixture

ELIGIBILITY:
Inclusion Criteria:

* Patients coming for elective and urgent coronary artery bypass (CABG)-only surgery.

Exclusion Criteria:

* Patients with a history of regular opioid use.
* Patients with a history of chronic pain.
* Patients unable to provide consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-01-26 (Actual); Primary Completion 2023-04-28 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Pain with inspirometry at 24 hours after surgery | 24 hours after surgery
  Numerical Rating Scale (NRS) pain score from the sternotomy site during inspirometry. The VAS score is a scale from 0 to 10 where 0 is equivalent to "no pain" and 10 is equal to "the worst imaginable pain"

SECONDARY OUTCOMES:
Opioid consumption | 12, 24 and 48 hours after surgery
  Amount of opioid administered (mg of Dilaudid)
Amount of rescue analgesia administered | Total in the first 48 hours after surgery
  Amount of ketorolac or ketamine administered
Pain score at rest | 12, 24 and 48 hours after surgery
  Numerical Rating Scale (NRS) pain score from the sternotomy site during inspirometry. The VAS score is a scale from 0 to 10 where 0 is equivalent to "no pain" and 10 is equal to "the worst imaginable pain"
Pain score with inspirometry | 12 and 48 hours after surgery
  Numerical Rating Scale (NRS) pain score from the sternotomy site during inspirometry. The VAS score is a scale from 0 to 10 where 0 is equivalent to "no pain" and 10 is equal to "the worst imaginable pain"
Intensive Care Unit (ICU) Length of Stay | From surgery until discharge from the ICU, assessed from the date of surgery up until 6 months after the completion of the study
  Time spent in the intensive care unit after surgery (days)
Hospital Length of Stay | From the date of surgery up until discharge from hospital, followed from the date of surgery up until 6 months after the completion of the study
  Time spent in the hospital after surgery (days)
Inspirometry | 24 hours after surgery
  Volume inspired on inspirometry
Patient satisfaction with pain control | at 48 hours after surgery
  0 "extremely unsatisfied" to 10 "extremely satisfied"
Mobilization | From ICU arrival until first mobilization (approximately first 48 hours postoperatively)
  Time from ICU arrival to the first mobilization to a chair
Ambulation | From ICU arrival until first ambulation (approximately first 72 hours postoperatively)
  Time from ICU arrival to the first mobilization to a chair

OTHER OUTCOMES:
Presence of postoperative vomiting | first 48 hours after surgery
  Vomiting after surgery
Incidence of bradycardia | first 48 hours after surgery
  Heart rate less than 60 beats per minute
Incidence of hyperglycemia | first 48 hours after surgery
  Glucose greater than 10 millimoles/liter
Incidence of a pneumothorax | first 48 hours after surgery
  Pneumothorax identified on chest x-ray
Local anesthetic toxicity | first 48 hours after surgery
  Local anesthetic toxicity, as diagnosed clinically
Postoperative Delirium | first 48 hours after surgery
  Delirium as defined by the "Confusion assessment method for the ICU" (CAM-ICU)
Narcotic prescription on discharge | Upon discharge from hospital after surgery (approximately 1 week after surgery)
  Having a narcotic prescription on discharge
Sternal pain at 3 months | Three months after the day of surgery
  Persistent pain at the sternum
Local anesthetic spread | Immediately as intervention is performed
  Number of levels of spread of local anesthetic, as identified by ultrasound

CONTACTS AND LOCATIONS:
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Cameron MJ, Long J, Yang SS, Kardash K. How Many Patients Are Needed to Detect a Difference in Pain With Parasternal Blocks? Anesth Analg. 2025 Jul 1;141(1):210-211. doi: 10.1213/ANE.0000000000007355. Epub 2024 Dec 17. No abstract available. PMID 39689005